CLINICAL TRIAL: NCT07080229
Title: The Effect of Intranasal Dexmedetomidine Compared to Placebo on Blood Pressure in Elderly Hypertensive Patients Undergoing Cataract Surgery: A Double-Blind Randomized Controlled Trial
Brief Title: Intranasal Dexmedetomidine on Blood Pressure in Elderly Hypertensive Patients Undergoing Cataract Surgery
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Principal Investigator, Mohammad E Salama, MD, Principal investigator, Suez Canal University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 5989#
Record Dates: First submitted 2025-07-14; First posted 2025-07-23 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Cataract; Hypertension
Keywords: Cataract; Hypertension; Intranasal Dexmedetomidine; Elderly
MeSH Terms: conditions — Cataract; Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexmedetomidine group (Study group) (Active Comparator): In this group, Dexmedetomidine (1 mcg/kg ideal body weight) will be administered intranasally 30 minutes before surgery.
  Interventions: Drug: Intranasal dexmedetomidine
- Placebo group (Control group) (Placebo Comparator): In this group, Normal Saline will be administered intranasally 30 minutes before surgery.
  Interventions: Drug: Intranasal normal saline

INTERVENTIONS:
Drug: Intranasal dexmedetomidine — Intranasal dexmedetomidine (1 mcg/kg ideal body weight) will be diluted to a total volume of 1 ml and will be administered via a mucosal atomization device (MAD) 30 minutes before surgery. The dose will be divided evenly, with 0.5 mL sprayed into each nostril while the patient is in a semi-recumbent position.
  Arms: Dexmedetomidine group (Study group)
Drug: Intranasal normal saline — Intranasal normal saline (1 ml) will be administered via mucosal atomization device (MAD) 30 minutes before surgery. The dose will be divided evenly, with 0.5 mL sprayed into each nostril while the patient is in a semi-recumbent position.
  Arms: Placebo group (Control group)

SUMMARY:
Cataract surgery in elderly patients with controlled hypertension carries a risk of hemodynamic instability, particularly fluctuations in mean arterial blood pressure (MAP). Dexmedetomidine, a selective α2-adrenergic agonist, offers hemodynamic stabilization and sedation when administered intranasally and provides a simple and non-invasive premedication option.

This study evaluates the effects of intranasal dexmedetomidine on perioperative mean arterial blood pressure in patients undergoing cataract surgeries.

Research Question:

Does intranasal dexmedetomidine premedication control blood pressure in elderly hypertensive patients undergoing cataract surgery?

Research Hypothesis:

Intranasal dexmedetomidine significantly reduces MAP and improves secondary outcomes compared to placebo.

Primary Objective: To evaluate the efficacy of intranasal Dexmedetomidine as a premedication to control hypertension in elderly patients scheduled for cataract surgery.

Secondary Objectives: 1. To assess surgery cancellation rates. 2. To evaluate satisfaction levels among patients, anesthesiologists, and surgeons using the Modified Observer's assessment of alertness/sedation scale (MOAA/S). 3- To evaluate the effect of intranasal dexmedetomidine on HR multiple readings starting from preoperative hold area till 2 hours postoperatively.

This randomized, double-blinded clinical trial will include 126 elderly hypertensive patients (≥65 years) undergoing cataract surgery under local anesthesia. Inclusion Criteria will consist of patients aged ≥65 years, ASA II or III, stage 2 hypertension as per ACC / AHA guidelines (SBP>140 and DBP> 90 mmHg), undergoing elective cataract surgery under local anesthesia. Exclusion Criteria will include allergy or contraindication to dexmedetomidine, significant baseline bradycardia (<50 bpm) or arrhythmia, use of sedative or anxiolytic medications, history of severe hepatic, renal, or cerebrovascular disease. Participants will be randomly assigned to receive either intranasal dexmedetomidine (1 mcg/kg ideal body weight) or a placebo (normal saline) 30 minutes before surgery. MAP, HR, and SpO₂ will be recorded at multiple perioperative intervals, and surgical cancellation rates, satisfaction levels will be noted, surgical duration, and hospital stay will be documented.

DETAILED DESCRIPTION:
Intranasal Administration Technique:

1. Intranasal dexmedetomidine (1 mcg/kg ideal body weight) will be diluted to a total volume of 1 ml.
2. A mucosal atomization device (MAD) will be used for administration.
3. The dose will be divided evenly, with 0.5 mL sprayed into each nostril while the patient is in a semi-recumbent position.
4. The control group will receive an equivalent volume of 0.9% saline using the same method.

Local Anesthesia A peribulbar block will be administered with a mixture of lidocaine 2% and bupivacaine 0.5% (total volume: 5 mL).

The block will be performed under aseptic conditions by an experienced anesthesiologist.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥65 years.
2. Patients who will have stage 2 hypertension as per ACC/AHA guidelines (Systolic BP > 140 and Diastolic BP> 90 mmHg)
3. Elective cataract surgery under local anesthesia.
4. American Society of Anesthesiologists (ASA) physical status II or III.

Exclusion Criteria:

1. Allergy or contraindication to dexmedetomidine.
2. Significant baseline bradycardia (<50 bpm) or arrhythmias.
3. Use of sedative or anxiolytic medications.
4. History of severe hepatic, renal, or cerebrovascular diseases.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2025-07-16 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Mean arterial blood pressure (MAP) | From preoperative baseline until 2 hours postoperatively
  Mean arterial blood pressure (MAP), measured in mmHg, will be recorded in both groups at the following time points:
  * Preoperative baseline
  * Every 5 minutes after intranasal drug administration
  * Intraoperative baseline
  * Immediately after peribulbar block
  * Every 5 minutes after the block until the end of the surgery
  * Every 15 minutes postoperatively until discharge

SECONDARY OUTCOMES:
Surgical cancellation rate | From the preoperative period until completion or cancellation of the surgery
  The number and percentage of cases in each group in which cataract surgery will be cancelled due to uncontrolled blood pressure, inadequate sedation, patient anxiety, or any other reason
Satisfaction score of patient, anesthesiologist, and surgeon using the Modified Observer's Assessment of Alertness/Sedation Scale (MOAA/S). | From preoperative drug administration until 2 hours postoperatively
  Sedation will be evaluated using the MOAA/S scale at predefined time points:
  * Every 5 minutes after intranasal drug administration
  * Intraoperative baseline
  * Immediately after peribulbar block
  * Every 5 minutes after the block until the end of the surgery
  * Every 15 minutes postoperatively until discharge
  The MOAA/S is a scale from 0 to 5 assessing a subject's responsiveness to verbal and physical stimuli as follows:
  0: No response after painful stimuli
  1. Responds only after painful trapezius squeeze
  2. Responds only after mild prodding or shaking
  3. Responds only after name is called loudly and/or repeatedly
  4. Lethargic response to name spoken in normal tone
  5. Responds readily to name spoken in normal tone
Heart rate (HR) | From preoperative baseline until 2 hours postoperatively
  Heart rate (HR) will be recorded in both groups at the following time points:
  * Preoperative baseline
  * Every 5 minutes after intranasal drug administration
  * Intraoperative baseline
  * Immediately after peribulbar block
  * Every 5 minutes after the block until the end of the surgery
  * Every 15 minutes postoperatively until discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Suez Canal University Hospitals, Ismailia, Ismailia Governorate, Egypt

REFERENCES:
- [Background] Wang K, Wu M, Xu J, Wu C, Zhang B, Wang G, Ma D. Effects of dexmedetomidine on perioperative stress, inflammation, and immune function: systematic review and meta-analysis. Br J Anaesth. 2019 Dec;123(6):777-794. doi: 10.1016/j.bja.2019.07.027. Epub 2019 Oct 24. PMID 31668347
- [Background] Rawlins JM, Segree W. Suggestions for increased job satisfaction for doctors and for improved patient care. West Indian Med J. 1984 Jun;33(2):87-91. No abstract available. PMID 6485320
- [Background] Xu X, Cao Y, Wu Y, Ding M. Intranasal Dexmedetomidine in Elderly Patients (Aged > 65 Years) During Maxillofacial Surgery: Sedative Properties and Safety Analysis. J Oral Maxillofac Surg. 2022 Mar;80(3):443-455. doi: 10.1016/j.joms.2021.10.013. Epub 2021 Oct 30. PMID 34838503
- [Background] Li A, Yuen VM, Goulay-Dufay S, Sheng Y, Standing JF, Kwok PCL, Leung MKM, Leung AS, Wong ICK, Irwin MG. Pharmacokinetic and pharmacodynamic study of intranasal and intravenous dexmedetomidine. Br J Anaesth. 2018 May;120(5):960-968. doi: 10.1016/j.bja.2017.11.100. Epub 2018 Feb 2. PMID 29661413
- [Background] Fleisher LA, Fleischmann KE, Auerbach AD, Barnason SA, Beckman JA, Bozkurt B, Davila-Roman VG, Gerhard-Herman MD, Holly TA, Kane GC, Marine JE, Nelson MT, Spencer CC, Thompson A, Ting HH, Uretsky BF, Wijeysundera DN. 2014 ACC/AHA guideline on perioperative cardiovascular evaluation and management of patients undergoing noncardiac surgery: executive summary: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines. Circulation. 2014 Dec 9;130(24):2215-45. doi: 10.1161/CIR.0000000000000105. Epub 2014 Aug 1. No abstract available. PMID 25085962
- [Background] Fang R, Yu YF, Li EJ, Lv NX, Liu ZC, Zhou HG, Song XD. Global, regional, national burden and gender disparity of cataract: findings from the global burden of disease study 2019. BMC Public Health. 2022 Nov 12;22(1):2068. doi: 10.1186/s12889-022-14491-0. PMID 36369026